Study Title: Effect of bisphosphonate use on surgical weight loss associated bone loss in older adults

with morbid obesity (WEight loss with RISEdronate for bone health; WE RISE)

IRB00048310 NCT03411902 Date: 10/1/20

Principal Investigator, Co-investigator(s): Co-PIs: Kristen Beavers and Jamy Ard. Co-Is: Adolfo

Fernandez, Daniel Beavers, Ashley Weaver, and Laura Flores

Sponsor or Funding Source: Internal

## **Background, Rationale and Context**

### 1. Significance

- 1.A. Osteoporosis is a significant public health problem in older adults with obesity, which may be exacerbated with weight loss. Worldwide, one in three women and one in five men over the age of 50 will experience an osteoporotic fracture in their lifetimes, with prevalence highest among those who are overweight and obese. Osteoporosis-related fractures of the hip and spine are the leading causes of injury in older adults, compromising both quality and expectancy of life. Bone mineral density (BMD) is a strong predictor of future osteoporotic fracture, with observational data consistently linking weight loss in late life with loss of BMD and increased fracture risk, regardless of intentionality of weight loss or initial body weight. 3,4 This finding is echoed in the randomized controlled trial literature, where dietary-induced weight loss interventions of at least 6 months in duration are consistently associated with small, but significant, decreases in total hip BMD (on the order of 0.010-0.015 g/cm<sup>2</sup> and conferring a 10-15% increase in fracture risk).<sup>5</sup> Accordingly, greater weight loss exacerbates this decline in BMD and subsequent risk of fracture, <sup>6-8</sup> with meta-analytic data showing BMD at the hip and spine is reduced by 0.1 g/cm<sup>2</sup> in the year following bariatric surgery (yielding ~35% weight loss), 9 representing a 10% decline from pretreatment values, 10 times what is expected from lifestyle-based interventions, and similar in magnitude to what is seen in studies of unloading. Alarmingly, emerging long-term data suggest that bone loss continues in these patients even after weight stabilizes, 9,10 with deterioration seen up to 5 years postsurgery. 11 Thus, of mounting concern to clinicians and patients, despite well recognized improvements in body weight and cardiometabolic indices, collective evidence suggests bariatric surgery irreversibly increases skeletal fragility and fracture risk, providing impetus to identify effective strategies to minimize bone loss during active weight loss in these patients.
- **1.B.** Bisphosphonate use reduces osteoporotic fracture risk and may be effective in minimizing surgical weight loss associated bone loss. Several FDA-approved pharmacotherapeutic options for osteoporosis are available at this time, and include: antiresorptive agents (i.e., bisphosphonates), selective estrogen receptor modulators (i.e., raloxifene), and hormonal agents (i.e., estrogen, teraparatide). Bisphosphonates are the most commonly prescribed drug to treat osteoporosis, and act by inhibiting activity of osteoclast cells, thereby decreasing the rate of bone resorption. Among oral bisphosphonates, Alendronate and Risedronate have been shown to reduce the number of vertebral and hip fractures, with Risedronate associated with significantly lower incidence of gastric and esophageal ulcers than Alendronate. Ulcinical practice guidelines support the consideration of oral bisphosphonate use in bariatric surgery patients with osteoporosis (provided that concerns about absorption or potential anastomotic ulceration are obviated), but no studies have examined the efficacy of oral bisphosphonate use to prophylactically attenuate surgical weight loss associated bone loss. Because weight loss is associated with a significant increase in bone resorption, for the prophylactical in reducing long-term fracture risk in bariatric surgery patients.
- 1.C. Current evidence on the effect of surgical-induced weight loss on measures of bone health are limited to traditional BMD metrics, select procedures, and younger populations. Dual-energy x-ray absorptiometry (DXA) acquired areal (a)BMD is the primary metric by which osteoporosis is assessed. However, more than half of all fractures occur in persons without osteoporosis (defined by aBMD), <sup>18</sup> indicating aBMD alone cannot sufficiently quantify all future fracture risk. Furthermore, acquisition of aBMD in the context of obesity and weight loss is limited by methodological issues (e.g., influence of adipose tissue on aBMD measurement, overall reduction in precision). Increasingly, volumetric BMD (vBMD) obtained with quantitative computed tomography (CT) is used to complement DXA-acquired aBMD estimates, <sup>19</sup> as less concern exists about obesity and weight loss-induced measurement error. <sup>20</sup> Further, CT allows for assessment of additional parameters of bone quality, including structure and strength, which add to fracture risk predictive power. <sup>21–23</sup> In addition to CT-derived measures of bone

quality, integration of biomarkers of bone metabolism with skeletal imaging data provide an early and sensitive measure of bone remodeling, and positively correlate with BMD and fracture risk. <sup>24</sup>

Studies assessing the effect of bariatric surgery on bone quality are less numerous and consistent than DXA studies, 7,10-14 and most are limited to data collected following the Roux-en-Y gastric bypass (RYBG) procedure and at peripheral sites (i.e., radius and tibia). Recently, there has been a national shift away from RYGB procedures in favor of sleeve gastrectomy (SG; comprises 50% of surgical weight loss procedures performed at Wake Forest Weight Management Clinic [WMC]). 28 This may have important implications on bone health, as nutrient deficiencies and ulcerations are less likely with SG; however, little empirical evidence exists to guide clinical understanding. To our knowledge only one study, conducted in primarily young to middle-aged adults, has been published examining the effects of SG (and RYGB) gastrectomy on aBMD and vBMD. 29 Authors report losses of hip and spine aBMD and vBMD in both groups, with potentially greater hip losses experienced in the RYGB group; although, findings warrant replication, particularly in older adults as they are at elevated risk of fracture.

#### **Objectives**

The main objective of this pilot project is to determine the feasibility of recruiting, enrolling, treating, and following 24 older SG patients into a randomized controlled trial (RCT) examining the efficacy of bisphosphonate use (versus placebo) in the prevention of surgical weight loss associated loss of bone mass and quality.

### **Methods and Measures**

## Design and Setting

This pilot study is a RCT, involving 24 participants randomized to consume Risedronate or placebo capsules for 24 weeks, and then followed for an additional 6 months. Two in-person baseline assessment visits [baseline visit 1 (BV1), baseline visit 2 (BV2)] occurring 1-6 weeks prior to surgery, two in-person 6 month follow up assessment visits [follow up visit 1 (FV1) and follow up visit 2 (FV2)] occurring within 1 month of their last pill date, and two, in-person 12 month follow up legacy assessment visits (FV3 and FV4) occurring within 1.5 months of their surgical anniversary date, as well as monthly medication compliance reminders and adverse event reporting during the active intervention period via phone (see **Table 1**). The Wake Forest WMC, under the direction of Drs. Ard and Fernandez, will serve as a source of recruitment for potential study participants.

**Table 1.** Proposed Study Assessment Timeline.

| Location: | WFU | WFSM | WFU | WFU | WFSM | WFU | WFSM |
|---|---|---|---|---|---|---|---|
| Week/Month Number: | -6 to -3 | -3 to -1 | -1 to<br>+23 | Within 1 month following last pill date | | Within 1.5 months of<br>their surgery date<br>anniversary | |
| | BV1 | BV2 | INT | FV1 | FV2 | FV3 | FV4 |
| Informed Consent | X | | | | | | |
| Demographic Characteristics | X | | | | | | |
| Medical History/Medication Use | X | | X | | | | |
| BMD/FRAX Questionnaire | X | | | X | | X | |
| DXA Assessment (total body and regional BMD) | Х | | | X | | X | |
| CT Assessment (hip/spine vBMD and bone quality) | | X | | | X | | X |
| Fasting Blood Draw for | | X | | | X | | X |

| Biomarkers of bone turnover | | |
|-----------------------------------|---|---|
| Monthly Medication | | |
| Compliance reminders and | X | |
| Adverse Event Collection | | |
| Participation Satisfaction Survey | | X |

## Participant Recruitment and Subject Selection Criteria

All subjects planning a SG procedure will be approached during their pre-surgical evaluation for possible participation in the study. Phase I exclusion criteria will be evaluated by phone screen and include age <40 years, baseline weight >450 pounds (DXA limit), chronic anti-reflux treatment, history of medical disorders known to affect bone metabolism, use of bone-active medications, or a known allergy to Risedronate. Participants who are given Phase I clearance will be further evaluated by the study physician (Drs. Ard/Fernandez, Phase II clearance) for potential eligibility (see **Table 2**). Eligible participants will be referred onto the study coordinator to read/sign an IRB-approved informed consent prior to enrollment.

**Table 2.** Proposed Inclusion and Exclusion Criteria.

| Clearance | Criteria | Inclusion | Exclusion | Assessment |
|---|---|---|---|---|
| Phase I | Sleeve Gastrectomy | Yes | | Referred from WMC |
| | Age | 40-79 years | | Self-report |
| | Weight Status | | Weight greater than 450 lbs (DXA | Scale |
| | | | limit) | |
| | Medicationuse | | Regular use of growth hormones, ora | Medical Record |
| | | | steroids, or prescription osteoporosis | |
| | | | medications; known allergies to | |
| | | | bisphosphonates. Unstable gastric | |
| | | | reflux requiring 2 or more additional | |
| | | | doses per month of anti-reflux | |
| | D | W/:II: 4 | medication. | C-16 |
| | Research participation | Willing to provide informed consent; | Current participation in other research study; Unable to provide own | Self-report |
| | | agree to all study | transportation to study visits; unable | |
| | | procedures and | to position on scanner independently. | |
| | | assessments. | to position on scanner independently. | |
| Phase II | Physician Clearance | Study MD | Participant presents with clinical | Medical Record or |
| | | approves safe | contraindications (i.e. creatinine | study baseline DXA |
| | | participation. | clearance < 30, hypocalcemia, | scan |
| | | | osteoporosis, pregnancy, esophageal | |
| | | | abnormalities, increased risk of | |
| | | | ulceration or electrolyte | |
| | | | abnormalities) | |

#### Sample Size

Twenty-four patients will be recruited to participate, with 12 randomized to the Risedronate group and 12 randomized to the placebo group, blocking by gender. Because this pilot is focused on feasibility and gathering evidence to inform future studies, all analyses are exploratory rather than confirmatory.

#### **Interventions and Interactions**

Risedronate is a pyridinyl bisphosphonate with potent anti-resorptive activity<sup>30,31</sup> which was approved at the 150 mg monthly dose for the prevention and treatment of post-menopausal osteoporosis.<sup>32</sup> Subjects randomized to the Risedronate group will take a 150 mg capsule of oral Risedronate once every 4 weeks for 24 weeks (6 doses), beginning 1 week prior to surgery. One bottle containing 6 blinded capsules will be dispensed from the WFSM research pharmacy to each participant at the second baseline visit (BV2).

Participants will be instructed to follow label instructions for the proper method of medication intake to minimize GI discomfort (i.e., take medication with 6-8 oz of plain water, remain upright for the next 30 minutes, avoid taking vitamins, mineral supplements, or antacids at the same time). Supplemental calcium and vitamin D will be provided to participants as a part of their post-surgical care and participants will be asked to take these supplements at least 30 minutes after taking the study medication. Participants randomized to the placebo group will receive identical placebo capsules and follow the same dosing protocol as the active treatment group, with both participants and study staff blinded to treatment allocation. To aid in compliance and safety monitoring, participants will receive monthly phone reminders to take their medications and will be queried for potential pregnancy (if applicable) and any new adverse events. After completing the active intervention period, subjects will return for follow up testing (i.e. FV1, FV2) and then return to free living conditions. Because bone remodeling requires a minimum of 4-6 months and continues for at least 12 months, 3 subjects will be asked to return within the one month following their surgical date anniversary date for additional follow up testing (FV3, FV4) to examine intervention legacy effects.

#### Assessments

## DXA-Acquired Outcome Measures

All DXA-acquired outcome measures will be assessed at BV1 and FV1. If obtainable, total body composition as well as areal BMD of the total hip, femoral neck, lumbar spine and distal radius and Trabecular Bone Score of the lumbar spine will be determined by DXA (iDXA, GE Medical Systems, Madison, WI), housed within the Wake Forest University Department of Health and Exercise Science. All scans will be performed and analyzed in accordance with national recommendations by an International Society for Clinical Densitometry (ISCD) trained DXA technologist.

## CT-Acquired Outcome Measures

All CT-acquired outcome measures will be assessed at BV2 and FV2. Single-energy helical CT scans of the femurs and lumbar spine will be acquired on a Siemens SOMATOM Definition Flash dual source CT scanner, housed within the WFSM, Department of Radiology. The scan coverage for the lumbar spine will be from the top of L1 through the base of L5, and the bilateral femur scan will cover the region from the superior acetabulum to mid-femur. Both scans will be conducted at SFOV 50 cm, 120 KVp, 350 mA, 1 mm helical with a pitch of 1, and a gantry speed 0.8 second, standard reconstruction, with secondary reconstruction set at 0.625 mm thick, bone algorithm. A 5-port bone mineral calibration phantom (Mindways Software, Inc., Austin, TX) will be imaged in every scan to allow for measurement of vBMD.<sup>34</sup> Quality assurance and processing of CT images for cortical thickness and finite element derived strength estimates will be performed according to published methodology by Dr. Weaver (select examples in **Figure 1**).<sup>35,36</sup>



**Figure 1. A)** Exemplar lumbar CT with Mindways phantom. **B)** Lumbar and hip vBMD measurement in QCT Pro<sup>TM</sup>. **C)** Older male from experienced cortical thinning relative to baseline (left) following 6.8% weight loss over 18 months (right).

## Biomarkers of Bone Turnover

Blood samples will be collected at BV2 and FV2 via venipuncture after an overnight fast (of ≥10 hours) and abstinence from physical activity for the previous 24 hours. After centrifugation for 20 minutes at

4°C, aliquots of serum will be stored at -70°C. Analyses of a bone formation marker (Procollagen Type 1 N-Terminal Propeptide, P1NP), and a bone resorption marker (C-Terminal Telopeptide of Type 1 Collagen, CTX) will be performed, by technicians in the ELISA Core laboratory using commercially available ELISAs (Neo Scientific, Cambridge, MA) as done previously.<sup>37</sup>

#### Baseline and Covariate Measures

Self-reported demographic information (i.e., age, gender, ethnicity, socioeconomic status) will be assessed at BV1. Participants will be queried at BV1 and FV1 on medical information relevant to assess 10-year major osteoporotic and hip fracture risk using the FRAX tool. <sup>38</sup> We will also record medication use by asking participants to bring in all medications (including nutritional supplements) and electronic medical records will be reviewed to assess co-morbid conditions.

## **Analytic Plan**

This pilot is focused on feasibility and gathering evidence to inform future studies; thus, all analyses are considered exploratory rather than confirmatory. Baseline characteristics will be summarized using descriptive measures both overall and by gender at baseline. Feasibility will be based on retention of participants at follow-up visits. Follow-up treatment effect estimates at 6 and 12 months on bone metrics will yield means, standard deviations, and within-person correlations for use in power estimates for future clinical trials. Secondary analyses will examine change in bone metrics predicted by the magnitude of weight lost using linear regression models and adjusted for baseline values, as well as whether associations differ across demographic (i.e. gender, race) subgroups. Dr. Daniel Beavers will oversee all statistical analyses.

### **Human Subjects Protection**

### Subject Recruitment Methods

The WMC will serve as the source of recruitment for potential study participants. Based on 216 sleeve gastrectomy procedures performed in FY2016 (average age 44.5 years), we expect a total recruitment pool of 18 participants/month, of which we anticipate a 35% recruitment rate to our study. Thus, enrollment of 6 participants/month with a baseline assessment (occurring 3-6 weeks prior to surgery) and follow up assessment occurring in the month following their last pill date, will allow us to recruit 20-24 participants within the allotted time period. All subjects planning a SG procedure will be approached during their pre-surgical evaluation by the WMC Surgery Coordinator for possible participation in the study. Contact information interested participants will be referred to the study coordinator for phone screen, eligibility (see **Table 2**), and potential scheduling of BV1.

### Sources of Research Material

Participants will self-report personal information on paper survey forms including personal demographic data, race, health information, psychological, social, and study satisfaction data. Results will also be recorded in a computer database. Data from the paper forms will be entered into an electronic database on a computer workstation. All material and data will be obtained solely for research purposes.

#### Informed Consent

Interested participants who are eligible via a telephone screening interview, are invited to a baseline visit. The informed consent process will follow the procedures of the WFSM Institutional Review Board. The study interviewers explain the purpose, methods and extent of the study to prospective participants. The potential participant is asked to read the informed consent form and ask questions. The form is written in simple easy to understand language. We require study staff to review all of the key aspects of the study verbally with the potential participants. Staff are provided with a structured checklist for this purpose. Staff are then required to question potential participants to ascertain whether s/he has understood the information.

Potential participants who are illiterate or have impaired vision must have the consent read to them, followed by review of the checklist, opportunity for questions, and discussion. A copy of the signed and dated consent form will be given to participants, and the original document will be placed in subjects' individual study files, which will be stored in a secure location. In compliance with the Health Insurance Portability and Accountability Act (HIPAA) and the Standards for Privacy of Individually Identifiable Health Information of the Department of Health and Human Services, we will access personal health information only after obtaining informed consent.

According to the NIH and the Office of Human Research Protection (OHRP) guidelines, the informed consent will contain the following elements:

- 1. A statement that the study involves research.
- 2. An explanation of the purposes of the research.
- 3. The expected duration of the subject's participation.
- 4. A description of the procedures to be followed.
- 5. Identification of any procedures which are experimental.
- 6. A description of any reasonably foreseeable risks or discomforts to the subject.
- 7. A description of any benefits to the subject that may reasonably be expected from the research.
- 8. A disclosure of appropriate alternative procedures or courses of treatment, if any, that might be advantageous to the subject.
- 9. A statement describing the extent to which confidentiality of records identifying the subject will be maintained.
- 10. An explanation of whether any compensation and any medical treatments are available if a research-related injury occurs and, what these consist of, or where further information is obtained.
- 11. An explanation of whom to contact for answers to pertinent questions about the research and research subjects' rights, and whom to contact in the event of a research-related injury.
- 12. A statement that participation is voluntary, refusal to participate will involve no penalty or loss of benefits to which the subject is otherwise entitled, and the subject may discontinue participation at any time without penalty or loss of benefits, to which the subject is otherwise entitled.
- 13. Anticipated circumstances under which subject participation may be terminated by the investigator without regard to the subject's consent.
- 14. Any additional costs to the subject that may result from participation in the research.
- 15. The consequences of a subject's decision to withdraw from the research and procedures for orderly termination of participation by the subject.
- 16. A statement that significant new findings developed during the course of the research, which may relate to the subject's willingness to continue participation, will be provided to the subject.
- 17. The approximate number of subjects involved in the study.

#### Potential Risks

There are inherent potential risks to human subjects who participate in any research study and the potential risks to study participants in this study are listed below. Any injuries or illnesses (severe adverse events) during the course of a participant's enrollment in the study will be monitored regularly at monthly intervention sessions. A health risk of the study testing may be discovery of osteoporosis at during the DXA scan. Subjects who are identified as having hip or spine T-score value(s) of ≥-2.5 at baseline will be excluded from study participation. Participants identified as osteoporotic at any DXA assessment will be offered referral to a bone evaluation clinic. Health risks of the intervention include rare, but serious, side effects from taking Risedronate, including chest pain, difficulty or pain when swallowing, pain or burning under the ribs or in the back, new or worsening heartburn, severe or ongoing indigestion, severe joint, bone, or muscle pain, new or unusual pain in the thigh or hip, or jaw pain, numbness, or swelling. Less serious side effects may include mild stomach pain or upset stomach, flu-like symptoms, muscle pain, diarrhea, constipation, mild joint or back pain, or headache. Health risks of the assessment procedures include exposure to radiation from the DXA and CT scans. The amount of radiation that participants will

receive from these procedures is equivalent to a uniform whole body dose of 1449 mrem, or 29% of the yearly radiation exposure limit allowed for a radiation worker (5000 mrem).

### Safety Measures During the Intervention and Assessments

To control risk of further bone loss, persons identified as having osteoporosis will be excluded from study participation. To minimize potential risk of GI irritation, persons with a prior history of severe reflux will be excluded from study participation and all active participants will be instructed to take the medication following manufacturer recommendations (i.e., take the medication with 6-8 oz of plain water and remain upright for the next 30 minutes). To minimize assessment associated risk, all study assessments will be conducted by trained and certified staff. Safety precautions will be taken during all testing by applying standardized stopping criteria. If the participant reports pain, tightness or pressure in the chest, feeling faint, lightheaded or dizzy, or any other medical problems, the test will be stopped. When there are medically relevant findings, the participant will be told the cause for concern, and may be advised to consult his or her physician. If given permission by the participant, a letter will be sent to her primary care physician stating the concern. Because of the potential for pregnancy in some participants during the study, urinary pregnancy tests will be administered before each DXA/CT assessment, and all women of childbearing potential will be provided with monthly pregnancy tests, upon request. Should pregnancy be detected, participants will discontinue the intervention immediately and will not complete follow up DXA or CT assessments. However, because sleeve gastrectomy patients are advised not to become pregnant at least 12 months following their surgery, the estimated pregnancy risk is slight.

### Confidentiality and Privacy

Data will be used only in aggregate and no identifying characteristics of individuals will be published or presented. Results of testing will be sent to participant's private physicians if participants agree to this. Confidentiality of data is maintained by using research identification numbers which uniquely identify each individual. The information collected from participants in this study has a low potential for abuse because the data does not address sensitive issues. Nevertheless, appropriate measures are taken to prevent unauthorized use of study information. Data other than demographic information do not use names as an identifier. The research ID number is used. The research records are kept in locked cabinets in the Department of Health and Exercise Science, WFU. The files matching the participants' names and demographic information with the research ID numbers are kept in a separate room and locked file that uses a different key from that of all other files. Files may not be obtained from the research unit by persons other than research personnel, who are asked to sign a document agreeing to maintain the confidentiality of the information. After the study is completed, the local data will be stored with other completed research studies in a secured storage area.

### Data and Safety Monitoring

The Co-PIs (Drs. Kristen Beavers and Jamy Ard) will be responsible for the overall monitoring of the data and safety of study participants. The Co-PIs will be assisted by other members of the study staff.

# Reporting of Unanticipated Problems, Adverse Events or Deviations

Any unanticipated problems, serious and unexpected adverse events, deviations or protocol changes will be promptly reported by the Co-PIs or designated member of the research team to the IRB and sponsor or appropriate government agency if appropriate.

## References

1. Facts and Statistics | International Osteoporosis Foundation [Internet]. [cited 2017 Mar 29]. Available from: https://www.iofbonehealth.org/facts-statistics

- 2. Nielson CM, Srikanth P, Orwoll ES. Obesity and fracture in men and women: an epidemiologic perspective. J Bone Miner Res. 2012 Jan;27(1):1–10. PMID: 23348758
- 3. Ensrud KE, Ewing SK, Stone KL, Cauley JA, Bowman PJ, Cummings SR. Intentional and unintentional weight loss increase bone loss and hip fracture risk in older women. J Am Geriatr Soc. 2003 Dec;51(12):1740–1747. PMID: 14687352
- 4. Shapses SA, Sukumar D. Bone metabolism in obesity and weight loss. Annu Rev Nutr. 2012 Aug 21;32(1):287–309. PMID: 22809104
- 5. Zibellini J, Seimon RV, Lee CM, Gibson AA, Hsu MS, Shapses SA, Nguyen TV, Sainsbury A. Does diet-induced weight loss lead to bone loss in overweight or obese adults? A systematic review and meta-analysis of clinical trials. J Bone Miner Res. 2015 Dec 1;30(12):2168–2178. PMID: 26012544
- 6. Lu C-W, Chang Y-K, Chang H-H, Kuo C-S, Huang C-T, Hsu C-C, Huang K-C. Fracture Risk After Bariatric Surgery: A 12-Year Nationwide Cohort Study. Medicine (Baltimore). 2015 Dec;94(48):e2087. PMCID: PMC4674195
- 7. Nakamura KM, Haglind EGC, Clowes JA, Achenbach SJ, Atkinson EJ, Melton LJ, Kennel KA. Fracture risk following bariatric surgery: a population-based study. Osteoporos Int J Establ Result Coop Eur Found Osteoporos Natl Osteoporos Found USA. 2014 Jan;25(1):151–158. PMCID: PMC3939838
- 8. Yu EW, Lee MP, Landon JE, Lindeman KG, Kim SC. Fracture Risk After Bariatric Surgery: Rouxen-Y Gastric Bypass Versus Adjustable Gastric Banding. J Bone Miner Res Off J Am Soc Bone Miner Res. 2017 Jun;32(6):1229–1236. PMCID: PMC5466471
- 9. Shanbhogue VV, Støving RK, Frederiksen KH, Hanson S, Brixen K, Gram J, Jørgensen NR, Hansen S. Bone structural changes after gastric bypass surgery evaluated by HR-pQCT: a two-year longitudinal study. Eur J Endocrinol. 2017 Jun;176(6):685–693. PMCID: PMC5425940
- Yu EW, Bouxsein ML, Putman MS, Monis EL, Roy AE, Pratt JSA, Butsch WS, Finkelstein JS. Two-year changes in bone density after Roux-en-Y gastric bypass surgery. J Clin Endocrinol Metab. 2015 Apr;100(4):1452–1459. PMCID: PMC4399296
- 11. Gastric-Bypass Bone Loss Continues 5 Years Out [Internet]. Medscape. [cited 2017 Nov 21]. Available from: http://www.medscape.com/viewarticle/885861
- 12. Drake MT, Clarke BL, Khosla S. Bisphosphonates: mechanism of action and role in clinical practice. Mayo Clin Proc. 2008 Sep;83(9):1032–1045. PMCID: PMC2667901
- 13. Cranney A, Tugwell P, Adachi J, Weaver B, Zytaruk N, Papaioannou A, Robinson V, Shea B, Wells G, Guyatt G, Osteoporosis Methodology Group and The Osteoporosis Research Advisory Group. Meta-analyses of therapies for postmenopausal osteoporosis. III. Meta-analysis of risedronate for the treatment of postmenopausal osteoporosis. Endocr Rev. 2002 Aug;23(4):517–523. PMID: 12202466
- 14. Lanza FL, Hunt RH, Thomson AB, Provenza JM, Blank MA. Endoscopic comparison of esophageal and gastroduodenal effects of risedronate and alendronate in postmenopausal women. Gastroenterology. 2000 Sep;119(3):631–638. PMID: 10982755

- 15. Mechanick JI, Youdim A, Jones DB, Garvey WT, Hurley DL, McMahon MM, Heinberg LJ, Kushner R, Adams TD, Shikora S, Dixon JB, Brethauer S, American Association of Clinical Endocrinologists, Obesity Society, American Society for Metabolic & Bariatric Surgery. Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, The Obesity Society, and American Society for Metabolic & Bariatric Surgery. Obes Silver Spring Md. 2013 Mar;21 Suppl 1:S1-27. PMCID: PMC4142593
- 16. Villareal DT, Fontana L, Das SK, Redman L, Smith SR, Saltzman E, Bales C, Rochon J, Pieper C, Huang M, Lewis M, Schwartz AV, CALERIE Study Group. Effect of two-year caloric restriction on bone metabolism and bone mineral density in non-obese younger adults: a randomized clinical trial. J Bone Miner Res. 2016 Jan;31(1):40–51. PMID: 26332798
- 17. Crawford MR, Pham N, Khan L, Bena JF, Schauer PR, Kashyap SR. Increased bone turnover in type 2 diabetes patients randomized to bariatric surgery vs. medical therapy at 5 years. Endocr Pract Off J Am Coll Endocrinol Am Assoc Clin Endocrinol. 2017 Nov 16; PMID: 29144812
- 18. Nguyen ND, Eisman JA, Center JR, Nguyen TV. Risk factors for fracture in nonosteoporotic men and women. J Clin Endocrinol Metab. 2007 Mar;92(3):955–962. PMID: 17164302
- 19. Engelke K, Libanati C, Fuerst T, Zysset P, Genant HK. Advanced CT based In Vivo Methods for the Assessment of Bone Density, Structure, and Strength. Curr Osteoporos Rep. 2013 May 28;(1544-2241 (Electronic)). PMID: 23712690
- 20. Yu EW, Bouxsein M, Roy AE, Baldwin C, Cange A, Neer RM, Kaplan LM, Finkelstein JS. Bone loss after bariatric surgery: Discordant results between DXA and QCT bone density. J Bone Min Res. 2013 Aug 8;(1523-4681 (Electronic)). PMID: 23929784
- 21. Engelke K, Lang T, Khosla S, Qin L, Zysset P, Leslie WD, Shepherd JA, Schousboe JT. Clinical use of quantitative computed tomography (qct) of the hip in the management of osteoporosis in adults: the 2015 ISCD official positions-part I. J Clin Densitom. 2015 Sep;18(3):338–358. PMID: 26277851
- 22. Shepherd JA, Schousboe JT, Broy SB, Engelke K, Leslie WD. Executive Summary of the 2015 ISCD Position Development Conference on Advanced Measures From DXA and QCT: Fracture Prediction Beyond BMD. J Clin Densitom. 2015 Jul;18(3):274–86.
- 23. Zysset P, Qin L, Lang T, Khosla S, Leslie WD, Shepherd JA, Schousboe JT, Engelke K. Clinical use of quantitative computed tomography-based finite element analysis of the hip and spine in the management of osteoporosis in adults: the 2015 ISCD official positions-part II. J Clin Densitom. 2015 Sep;18(3):359–392. PMID: 26277852
- Vasikaran S, Eastell R, Bruyere O, Foldes AJ, Garnero P, Griesmacher A, McClung M, Morris HA, Silverman S, Trenti T, Wahl DA, Cooper C, Kanis JA, Group I-IBMSW. Markers of bone turnover for the prediction of fracture risk and monitoring of osteoporosis treatment: a need for international reference standards. Osteoporos Int. 2011 Feb;22(2):391–420. PMID: 21605012
- 25. Lima TP, Nicoletti CF, Marchini JS, Junior WS, Nonino CB. Effect of weight loss on bone mineral density determined by ultrasound of phalanges in obese women after Roux-en-y gastric bypass: conflicting results with dual-energy X-ray absorptiometry. J Clin Densitom Off J Int Soc Clin Densitom. 2014 Dec;17(4):473–478. PMID: 25443227

- 26. Frederiksen KD, Hanson S, Hansen S, Brixen K, Gram J, Jørgensen NR, Støving RK. Bone Structural Changes and Estimated Strength After Gastric Bypass Surgery Evaluated by HR-pQCT. Calcif Tissue Int. 2016 Mar;98(3):253–262. PMID: 26661530
- 27. Scibora LM, Buchwald H, Petit MA, Hughes J, Ikramuddin S. Bone strength is preserved following bariatric surgery. Obes Surg. 2015 Feb;25(2):263–270. PMID: 24972685
- 28. Estimate of Bariatric Surgery Numbers, 2011-2015 [Internet]. American Society for Metabolic and Bariatric Surgery. 2016 [cited 2017 Sep 8]. Available from: https://asmbs.org/resources/estimate-of-bariatric-surgery-numbers
- 29. Bredella MA, Greenblatt LB, Eajazi A, Torriani M, Yu EW. Effects of Roux-en-Y gastric bypass and sleeve gastrectomy on bone mineral density and marrow adipose tissue. Bone. 2017 Feb;95:85–90. PMCID: PMC5222731
- 30. McClung MR, Benhamou C-L, Man Z, Tlustochowicz W, Zanchetta JR, Eusebio R, Balske AM, Matzkin E, Olszynski WP, Recker R, Delmas PD. A novel monthly dosing regimen of risedronate for the treatment of postmenopausal osteoporosis: 2-year data. Calcif Tissue Int. 2013 Jan;92(1):59–67. PMCID: PMC3528955
- 31. Fogelman I, Ribot C, Smith R, Ethgen D, Sod E, Reginster JY. Risedronate reverses bone loss in postmenopausal women with low bone mass: results from a multinational, double-blind, placebo-controlled trial. BMD-MN Study Group. J Clin Endocrinol Metab. 2000 May;85(5):1895–1900. PMID: 10843171
- 32. Drug Approval Package: Actonel (Risedronate Sodium) NDA# 20-835 [Internet]. [cited 2017 Nov 27]. Available from: https://www.accessdata.fda.gov/drugsatfda\_docs/nda/98/20835\_Actonel.cfm
- 33. Heaney RP. The bone-remodeling transient: implications for the interpretation of clinical studies of bone mass change. J Bone Min Res. 1994 Oct;9(10):1515–1523.
- 34. Weaver AA, Beavers KM, Hightower RC, Lynch SK, Miller AN, Stitzel JD. Lumbar bone mineral density phantomless computed tomography measurements and correlation with age and fracture incidence. Traffic Inj Prev. 2015;16 Suppl 2:S153-160. PMID: 26436225
- 35. Okoukoni C, Randolph DM, McTyre ER, Kwok A, Weaver AA, Blackstock AW, Munley MT, Willey JS. Early dose-dependent cortical thinning of the femoral neck in anal cancer patients treated with pelvic radiation therapy. Bone. 2017 Jan;94:84–89. PMID: 27780791
- 36. Schoell SL, Weaver AA, Urban JE, Jones DA, Stitzel JD, Hwang E, Reed MP, Rupp JD, Hu J. Development and validation of an older occupant finite element model of a mid-sized male for investigation of age-related injury risk. Stapp Car Crash J. 2015 Nov;59:359–383. PMID: 26660751
- 37. Kelleher JL, Beavers DP, Henderson RM, Yow D, Crotts C, Kiel J, Nicklas BJ, Beavers KM. Weighted Vest Use during Dietary Weight Loss on Bone Health in Older Adults with Obesity. J Osteoporos Phys Act. 2017;5(4). PMCID: PMC5788462
- 38. Watts NB, Lewiecki EM, Miller PD, Baim S. National Osteoporosis Foundation 2008 clinician's guide to prevention and treatment of osteoporosis and the world health organization fracture risk assessment tool (FRAX): what they mean to the bone densitometrist and bone technologist. J Clin Densitom. 2008 Dec;11(4):473–477. PMID: 18562228